CLINICAL TRIAL: NCT03880695
Title: Anlotinib Hydrochloride Combined With Liposomal Doxorubicin in the Treatment of Locally Advanced or Metastatic Soft Tissue Sarcoma : a One-arm, Multi-center, Prospective Clinical Trial (ALTER-S001)
Brief Title: Anlotinib Hydrochloride Combined With Liposomal Doxorubicin in the Treatment of Locally Advanced or Metastatic Soft Tissue Sarcoma
Acronym: ALTER-S001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Peking University Cancer Hospital & Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other); The First Hospital of Jilin University (Other); Hunan Cancer Hospital (Other); Ruijin Hospital (Other); Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, GUO WEI, Principal Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018PHD008-01
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+ Liposomal Doxorubicin (Experimental): Anlotinib Hydrochloride Combined With Liposomal Doxorubicin Liposomal Doxorubicin 50mg/m2 Day 1 every-3-weeks (Q3W) and Anlotinib 12mg QD po at Day 8-21 Q3W and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent. Dose reductions/modifications will be applied as indicated by toxicities and/or patient tolerance.
  Interventions: Drug: Anlotinib+ Liposomal Doxorubicin

INTERVENTIONS:
Drug: Anlotinib+ Liposomal Doxorubicin — Anlotinib : 12 mg, qd, po day 8-21 every 3 weeks Liposomal Doxorubicin: 50 mg/m2, day 1 every 3 weeks
  Other Names: Anlotinib+ LPD

SUMMARY:
The investigators explored the activity of anlotinib combined with Liposomal Doxorubicin in patients with Locally Advanced or Metastatic Soft Tissue Sarcoma

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form prior to patient entry;
* ≥ 14 years of age , regardless of gender；ECOG :0-1;Expected Survival Time: Over 3 months;
* Histologically confirmed diagnosis of un-resectable or recurrent metastatic soft tissue sarcoma, such as: leiomyosarcoma, synovial sarcoma, undifferentiated pleomorphic sarcoma, liposarcoma , angiosarcoma, alveolar soft tissue sarcoma, and other sarcomas. The following histologies are excluded: embryonic rhabdomyosarcoma, chondrosarcoma, osteosarcoma, gastrointestinal stromal tumor and Ewing sarcoma/primary neuroectodermal tumor.
* Previously without anthracyclines or other anti-tumor drugs
* Evaluable disease by imaging or physical exam or measurable disease defined as at least one lesion that can be accurately measured according to RECIST version 1.1.
* Normal main organs function as defined below: Hemoglobin (Hb) ≥ 80g / L, Neutrophils (ANC) ≥ 1.5 × 10^9 / L, Platelet count (PLT) ≥ 80 × 10^9 / L, Serum creatinine (Cr) ≤ 1.5 × normal upper limit (ULN) or creatinine clearance (CCr) ≥ 60ml / min, Blood urea nitrogen (BUN) ≤ 2.5 × normal upper limit (ULN); Total bilirubin (TB) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; If accompanied by liver metastases, ALT and AST ≤ 5 × ULN Albumin (ALB) ≥ 25 g/L. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%)
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped.

Exclusion Criteria:

* Prior treatment with anlotinib or any other VEGFR tyrosine kinase inhibitor (such as sunitinib, sorafenib, bevacizumab, imatinib, famitinib, apatinib, regorafenib and other drugs).
* Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy, is planned for the first 4 weeks prior to enrollment or during the study. Radiation radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment.
* A history of other malignancy ≤ 3 years previous
* Known central nervous system metastases.
* Imaging (CT or MRI) shows tumor lesions from large vessels ≤ 5 mm, the tumor is very likely to invade the important blood vessels and cause fatal hemorrhage, or the formation of tumor thrombosis with large veins (iliac vessels, inferior vena cava, pulmonary veins, superior vena cava);
* The investigator judged that the presence of distinct pulmonary cavitary or necrotic tumors;
* Serosal effusion with clinical symptoms requiring surgical management (including hydrothorax and ascites pericardial effusion)
* With uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug treatment).
* Arrhythmias with grade II and above myocardial ischemia or myocardial infarction, poor control (including corrected QT interval(QTc) men ≥ 450 ms, women ≥ 470 ms).
* According to NYHA criteria, grade III to IV cardiac insufficiency, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%, myocardial infarction occurred within 6 months before enrollment, ≥ 2 congestive heart failure (New York Heart Association ( NYHA) rating ), uncontrolled angina, clinical pericardial disease, or electrocardiogram suggesting acute ischemia or active conduction system abnormalities.
* Uncontrolled comorbid diseases, including but not limited to: poorly controlled diabetes, persistent active infections, or mental illness or social condition that may affect a subject's adherence to the study.
* Patients with active hepatitis B or hepatitis C (hepatitis B: HBsAg-positive and hepatitis B virus(HBV) DNA ≥ 500 IU/mL; hepatitis C: hepatitis C virus(HCV) RNA-positive and abnormal liver function), or active infection requiring antimicrobial treatment (eg Treated with antibacterial drugs, antiviral drugs, antifungal drugs)
* Renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;
* Patients with seizures and need treatment
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time(APTT) > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy.
* Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin.
* Significant coughing blood in the 2 months before enrollment, or daily hemoptysis of 2.5ml or more.
* History of psychotropic substance abuse who are unable to quit or have a mental disorder.
* Tendencies of hereditary or acquired hemorrhagic and thrombotic (such as hemophilia patients, coagulopathy, thrombocytopenia, hypersplenism, etc.)
* Any major unhealed wound, ulcer, or fracture occurred in a patient who had undergone major surgery or trauma within 4 weeks prior to enrollment.
* Active period digestive ulcers.
* Cavity sinus or perforation occurred within 6 months.
* Participated in other anti-tumor clinical trials within 4 weeks.
* Received a potent CYP3A4 inhibitor (such as ketoconazole, itraconazole, erythromycin, and clarithromycin) within 7 days, or received a potent CYP3A4 inducer within 12 days prior to the study (eg. catarrh Treatment with imipramine, rifampicin and phenobarbital).
* Allergic reactions, hypersensitivity reactions or intolerance to anlotinib hydrochloride or its excipients.
* Pregnancy or lactation.
* The investigator believes that there are any conditions that may damage the subject or result in the subject not being able to meet or perform the research request.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Progress free survival (PFS) | each 42 days to evaluate up to intolerance the toxicity or PD (in first 24 weeks), each 84 days to evaluate up to intolerance the toxicity or PD (up to 24 months)
  Calculated from the date of treatment start until last follow-up or death, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
  Calculated from the date of treatment start until last follow-up or death, whichever comes first.
Objective Response Rate (ORR) | each 42 days to evaluate up to intolerance the toxicity or PD (in first 24 weeks), each 84 days to evaluate up to intolerance the toxicity or PD (up to 24 months)
  Overall objective response measured using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease Control Rate (DCR) | each 42 days to evaluate up to intolerance the toxicity or PD (in first 24 weeks), each 84 days to evaluate up to intolerance the toxicity or PD (up to 24 months)
  Disease Control Rate measured using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Quality of Life (QoL) | each 42 days to evaluate up to intolerance the toxicity or PD (in first 24 weeks), each 84 days to evaluate up to intolerance the toxicity or PD (up to 24 months)
  QoL is measured by the World Health Organization Quality of Life (WHOQOL-BREF)

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No